CLINICAL TRIAL: NCT03617432
Title: Chidamide With Cyclophosphamide, Doxorubicin, Vincristine, Prednisone and Etoposide for Peripheral T Cell Lymphoma Patients : a Prospective, Randomized Controlled, Open Label, Phase II Clinical Trial
Brief Title: Chidamide Combined With CHOPE Regimen for Peripheral T-cell Lymphoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Peking University International Hospital (Other); Shandong Tumor Hospital (Other); Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhu, Director of lymphoma department, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-T13
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Experimental Tumor
MeSH Terms: conditions — Neoplasms, Experimental | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Cyclophosphamide; Doxorubicin; Vincristine; Etoposide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group will be treated by Chidamide combined CHOPE (Cyclophosphamide, Doxorubicin, Vincristine, Prednisone and Etoposide ) regimen for 6 cycles.
  Interventions: Drug: Chidamide; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Etoposide; Drug: Prednisone
- Control group (Experimental): Control group will be treated by CHOPE (Cyclophosphamide, Doxorubicin, Vincristine, Prednisone and Etoposide ) regimen for 6 cycles.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Etoposide; Drug: Prednisone

INTERVENTIONS:
Drug: Chidamide — Chidamide 15mg orally BIW. Six cycles of therapy will be administered, and each cycle of treatment is 21 days.
  Other Names: epidaza
  Arms: Experimental group
Drug: Cyclophosphamide — Cyclophosphamide(750mg/m2) was administered intravenously on d1. Six cycles of therapy will be administered, and each cycle of treatment is 21 days.
Drug: Doxorubicin — Doxorubicin (50mg/m2)was administered intravenously on d1.Six cycles of therapy will be administered, and each cycle of treatment is 21 days.
Drug: Vincristine — Vincristine (1.4mg)was administered intravenously on d1.Six cycles of therapy will be administered, and each cycle of treatment is 21 days.
Drug: Etoposide — Etoposide (100mg/m2) was administered intravenously on d1,2,3.Six cycles of therapy will be administered, and each cycle of treatment is 21 days.
Drug: Prednisone — Prednisone (100mg)was administered by oral on d1-5.Six cycles of therapy will be administered, and each cycle of treatment is 21 days.

SUMMARY:
Chidamide With Cyclophosphamide, Doxorubicin, Vincristine, Prednisone and Etoposide for Peripheral T Cell Lymphoma Patients : a Prospective, Randomized Controlled, Open Label, Phase II Clinical Trial

DETAILED DESCRIPTION:
Chidamide，a novel histone deacetylase inhibitor has been approved for the treatment of relapsed or refractory peripheral T-cell lymphoma in China. The aim of this study was to observe the efficacy and safety of Chidamide With Cyclophosphamide, Doxorubicin, Vincristine, Prednisone and Etoposide for Peripheral T Cell Lymphoma Patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathology / cytology diagnosed as peripheral T cell lymphoma (PTCL) according to WHO 2016 classification criteria（NK/T cell lymphoma and ALK positive anaplastic large cell lymphoma excluded）including:Peripheral T-cell lymphoma, NOS，Angioimmunoblastic T-cell lymphoma，Anaplastic large-cell lymphoma, ALK negative，Enteropathy-associated T-cell lymphoma，Hepatosplenic T-cell lymphoma，Subcutaneous panniculitis T-cell lymphoma，Mycosis fungoides，Other T-cell lymphoma that investigators consider to be appropriate to be enrolled;
2. Patients have received CHOPE regimen for 2 cycles therapy and achieve PR or SD;
3. Patients should have at least one evaluable foci ( lymph nodes with diameter≥1.5cm, or evaluable skin foci);
4. Age 18-70 years, male or female;
5. ECOG performance status 0-2;
6. Absolute neutrophil count ≥1.5×109/L, platelet ≥75×109/L, Hb ≥ 90g/L;
7. ALT and serum creatinine <1.5 times of normal maximum;
8. Life expectancy no less than 3 months;
9. Willing to sign the Informed Consent Form.

Exclusion Criteria:

1. NK/T cell lymphoma or ALK positive anaplastic large cell lymphoma;
2. Female patients in lactation or pregnancy, Childbearing female or male patients unwilling to take contraceptive measures;
3. QTc elongation with clinical significance ( male> 450ms, female> 470ms), ventricular tachycardia, atrial fibrillation, cardiac conducting blockage, myocardial infarction within 1 year, congestive heart failure, symptomatic coronary heart disease that requires treatment;
4. Patients have undergone organ transplantation;
5. Patients received symptomatic treatment for bone marrow toxicity within 7 days prior to enrollment;
6. Patients with active hemorrhage;
7. Patients with or with history of thrombosis, embolism, cerebral hemorrhage, or cerebral infarction;
8. Patients with active infection or continuous fever within 14 days prior to enrollment;
9. Had major organ surgery within 6 weeks prior to enrollment;
10. Impaired liver function ( Total bilirubin > 1.5 times of normal maximum, ALT/AST> 2.5 times of normal maximum, for patients with infiltrative liver disease ALT/AST> 5 times of normal maximum), impaired renal function (serum creatinine> 1.5 times of normal maximum);
11. Patients with mental disorders or those do not have the ability to consent;
12. Patients with drug abuse, long term alcoholism that may impact the results of the trial;
13. Patients with invasion of central nervous system ;
14. Non-appropriate patients for the trial according to the judgment of the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
complete remission (CR）rate | up to 2 years
  The rate of patients who achieve complete remission after the treatment.

SECONDARY OUTCOMES:
objective response rate（ORR） | up to 2 years
  The total proportion of patients with complete response（CR）and partial response（PR）.
progression-free survival（PFS） | 2 years
  Time from treatment until disease progression or death.
overall survival（OS） | 2 years after the last patient's enrollment.
  From the date of inclusion to date of death, irrespective of any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No